CLINICAL TRIAL: NCT01196078
Title: A Phase II Randomized Trial of Erlotinib or Vinorelbine in Chemo-naive, Advanced, Non-Small-Cell Lung Cancer Patients Aged 70 Years or Older in Taiwan
Brief Title: A Study of Tarceva (Erlotinib) in Elderly Patients With Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML20322
Record Dates: First submitted 2010-09-03; First posted 2010-09-08 (Estimated); Results first posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-06

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride; Vinorelbine

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: erlotinib [Tarceva]
- 2 (Active Comparator)
  Interventions: Drug: vinorelbine

INTERVENTIONS:
Drug: erlotinib [Tarceva] — 150 mg, orally once a day for up to 6 cycles of 21 days each
  Arms: 1
Drug: vinorelbine — 60 mg/m2, orally on days 1 and 8 of cycle 1, 80 mg/m2 for the other cycles
  Arms: 2

SUMMARY:
This study will compare the efficacy and safety of Tarceva (erlotinib) and vinorelbine in chemo-naive elderly patients with advanced non-small cell lung cancer. Patients will be randomized to receive either Tarceva (150 mg po daily) or vinorelbine (60 mg/m2 on days 1 and 8 of cycle 1 and 80 mg/m2 for the other 21 days cycles). The anticipated time on study treatment is until disease progression.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, >=70 years of age
* Non-small cell lung cancer
* Naive to prior chemotherapy or specific immunotherapy
* Presence of at least 1 measurable lesion

Exclusion Criteria:

* Active non-controlled infection or disease
* CNS metastases
* Any other malignancies (other than adequately treated basal cell cancer of skin, or in situ cancer of the cervix)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 114 (Actual)
Dates: Start 2007-02; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (1):
- Taipei, Taiwan

RESULTS

PARTICIPANT FLOW:
Groups:
- Erlotinib: Participants received erlotinib 150 milligrams (mg), tablets, orally, once a day until disease progression, unacceptable toxicity, or participant withdrawal.
- Vinorelbine: Cycle 1 (21-day cycle): Participants received vinorelbine 60 milligrams per square meter (mg/m^2) orally on Days 1 and 8, followed by 1 week off.
  Cycles 2 and beyond (21-day-cycles): Participants received vinorelbine 80 mg/m^2 (in the absence of Grade 2 adverse events [AEs]) orally, on Days 1 and 8, followed by 1 week off. Treatment continued until disease progression, unacceptable toxicity, or participant withdrawal.
Period: Overall Study
Arm/Group | Erlotinib | Vinorelbine
Started | 57 | 57
Completed | 24 | 20
Not Completed | 33 | 37
Not completed — Withdrawal by Subject | 3 | 5
Not completed — Adverse Event | 4 | 4
Not completed — Protocol Violation | 2 | 1
Not completed — Lack of Efficacy | 17 | 23
Not completed — Lost to Follow-up | 1 | 0
Not completed — Death | 6 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: all randomized participants who received at least one dose of study medication.
Groups:
- Erlotinib: Participants received erlotinib 150 mg, tablets, orally, once a day until disease progression, unacceptable toxicity, or participant withdrawal.
- Vinorelbine: Cycle 1 (21-day cycle): Participants received vinorelbine 60 mg/m^2 orally on Days 1 and 8, followed by 1 week off.
  Cycles 2 and beyond (21-day-cycles): Participants received vinorelbine 80 mg/m^2 (in the absence of Grade 2 AEs) orally, on Days 1 and 8, followed by 1 week off. Treatment continued until disease progression, unacceptable toxicity, or participant withdrawal.
- Total: Total of all reporting groups
Arm/Group | Erlotinib | Vinorelbine | Total
Number analyzed (Participants) | 57 | 56 | 113
Age, Continuous [Mean (Standard Deviation); unit: years] | 78 (4.98) | 78 (5.32) | 78 (5.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 47 | 45 | 92

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Best Overall Response of Complete Response (CR) or Partial Response (PR)
Description: CR was defined as disappearance of all target lesions. PR was defined as at least a 30 percent (%) decrease in the sum of the longest diameter (LD) of target lesions, taking as reference the baseline sum LD. Participants experiencing either a CR or PR according to Response Evaluation Criteria in Solid Tumors (RECIST) were classified as responders. Participants with tumour assessment unevaluable were viewed as non-responders.
Time Frame: Screening, Day 1 of Cycles 3 and 5 and at End of treatment up to 1 year
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 57 | 56
percentage of participants | 22.81 | 8.93
Statistical Analysis 1: Comparison: Erlotinib vs Vinorelbine; Test type: Superiority or Other; p = 0.0388, Regression, Logistic — Between-treatment difference computed using logistic regression with treatment and multiple factors (gender, Eastern Cooperative Oncology Group [ECOG] status, histology status, and smoking status) as explanatory variables; Difference in Percentages = 13.88, 95% CI 2-sided [-0.22 to 26.19] — 95% confidence interval (CI) for the difference in tumor response rate determined using Hauck-Anderson approach

2. Secondary Outcome: Percentage of Participants Achieving Disease Control
Description: Disease control was defined as achieving a best overall response of CR, PR, or stable disease (SD) according to RECIST criteria. Participants with tumor assessment unevaluable were viewed as uncontrolled.
Time Frame: Screening, Day 1 of Cycles 3 and 5 and at End of treatment up to 1 year
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 57 | 56
percentage of participants | 71.93 | 57.14
Statistical Analysis 1: Comparison: Erlotinib vs Vinorelbine; Test type: Superiority or Other; p = 0.1061, Regression, Logistic — Between-treatment difference computed using logistic regression with treatment and multiple factors (gender, ECOG status, histology status, and smoking status) as explanatory variables; Difference in Percentages = 14.79, 95% CI 2-sided [-3.54 to 31.33] — 95% CI for the difference in the disease control rate determined using Hauck-Anderson approach

3. Secondary Outcome: Duration of Response Among Participants Who Achieved Either a CR or PR
Description: Duration of response was defined similarly for complete and partial responders. Complete response lasted from the date the complete response was first recorded to the date on which progressive disease was first noted or date of death. Partial response lasted from the date of partial response to the date of the first observation of progressive disease or date of death.
Time Frame: Screening, Day 1 of Cycles 3 and 5, every 4th cycle during post-study treatment, and every 3 cycles during follow-up
Population: ITT population; only participants with a response (CR or PR) were included in the analysis.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 13 | 5
months | 10.89 [5.48 to 22.23] | 8.75 [2.75 to NA] — Upper limit of the 95% CI could not be calculated because the duration of follow-up was too short to observe enough events for complete data estimation.
Statistical Analysis 1: Comparison: Erlotinib vs Vinorelbine; Test type: Superiority or Other; p = 0.9505, Log Rank

4. Secondary Outcome: Percentage of Participants With Disease Progression
Description: Progressive disease was defined using RECIST as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Day 1 of Cycles 1, 3, and 5 or first documentation of progressive disease or death
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 57 | 56
percentage of participants | 63.16 | 58.93

5. Secondary Outcome: Time to Disease Progression
Description: Time to disease progression was defined as the interval between the day of randomization and the first documentation of progressive disease or death.
Time Frame: Day 1 of Cycles 1, 3, and 5 or first documentation of progressive disease or death
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 57 | 56
months | 6.66 [4.43 to 9.05] | 3.87 [2.49 to 6.92]
Statistical Analysis 1: Comparison: Erlotinib vs Vinorelbine; Test type: Superiority or Other; p = 0.2314, Log Rank; Data were stratified by gender, ECOG status, histology status, and smoking status

6. Secondary Outcome: Overall Survival: Percentage of Participants With an Progressive Disease or Death
Description: Overall survival was defined as the time from the date of randomization to the date of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last dose and participants with no postbaseline information were censored at the time of randomization. Progressive disease was defined per RECIST as at least a 20% increase in the sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Day 1 of Cycles 1 through 6 to date of death or date of last follow-up assessment
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 57 | 56
percentage of participants | 56.14 | 48.21

7. Secondary Outcome: Overall Survival: Time to Event
Description: Overall survival was defined as the time from the date of randomization to the date of death. Participants who were alive at the time of the analysis were censored at the date of the last follow-up assessment. Participants without follow-up assessment were censored at the day of last dose and participants with no post baseline information were censored at the time of randomization. Overall median time to event was assessed for the population that experienced an event.
Time Frame: Day 1 of Cycles 1 through 6 to date of death or date of last follow-up assessment
Population: ITT population
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 57 | 56
months | 11.21 [6.79 to 19.57] | 10.36 [7.67 to NA] — Upper limit of the 95% CI could not be calculated because the duration of follow-up was too short to observe enough events for complete data estimation.
Statistical Analysis 1: Comparison: Erlotinib vs Vinorelbine; Test type: Superiority or Other; p = 0.9894, Log Rank; Data were stratified by gender, ECOG status, histology status, and smoking status

8. Secondary Outcome: Quality of Life as Measured by the Functional Assessment of Cancer Therapy (FACT) Questionnaire
Description: The FACT Questionnaire contains 4 general and 1 lung cancer symptom-specific subscale, including Physical Well-Being (PWB), Social/family Well-Being (SWB), Emotional Well-Being (EWB), Functional Well-Being (FWB), and the 8-item Lung Cancer Subscale (LCS) that assess symptoms commonly reported by participants with lung cancer. Each subscale was assessed by a five-point scale from 0 (not at all) to 4 (very much) to determine the quality of life. PWB, SWB and FWB scores ranged from 0-28 and EWB scores ranged from 0-24. LCS scores ranged from 0-36. For subscales of FWB and SWB, questionnaires of EWB, and additional concerns questions, the higher score represented 'Improved'. For other subscales and questionnaires, the higher score represented 'Worsened'. Missing data were replaced by the valid post-baseline assessment before. The FACT-L score ranges from 0 to 136, with higher scores indicating better quality of life.
Time Frame: Baseline and Day 1 of Cycles 2, 3, 4, 5, 6 and End of study
Population: Safety Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 57 | 55
units on a scale
  PWB, Baseline (n=56,53) | 6.8 (4.0) | 6.2 (3.7)
  PWB, Cycle 2 (n=52,42) | 8.1 (3.7) | 7.5 (4.4)
  PWB, Cycle 3 (n=41,28) | 8.9 (4.3) | 5.7 (4.2)
  PWB, Cycle 4 (n=37,28) | 9.4 (4.0) | 7.8 (6.1)
  PWB, Cycle 5 (n=30,22) | 8.8 (4.3) | 7.7 (5.5)
  PWB, Cycle 6 (n=25,20) | 9.3 (5.0) | 6.4 (5.5)
  PWB, End of Study (n=52,48) | 10.8 (5.2) | 7.8 (4.5)
  SWB, Baseline (n=55,53) | 15.9 (6.3) | 15.2 (6.8)
  SWB, Cycle 2 (n=52,40) | 15.5 (6.7) | 14.7 (7.2)
  SWB, Cycle 3 (n=42,30) | 16.0 (6.9) | 16.5 (6.8)
  SWB, Cycle 4 (n=37,27) | 15.9 (7.0) | 16.1 (7.1)
  SWB, Cycle 5 (n=28,21) | 15.7 (7.0) | 15.1 (7.7)
  SWB, Cycle 6 (n=26,18) | 15.2 (7.8) | 17.4 (7.1)
  SWB, End of Study (n=52,47) | 14.4 (7.1) | 14.3 (7.6)
  EWB, Baseline (n=57,55) | 7.8 (3.7) | 6.5 (3.4)
  EWB, Cycle 2 (n=52,43) | 6.7 (3.8) | 5.9 (3.2)
  EWB, Cycle 3 (n=42,29) | 6.4 (3.5) | 5.6 (2.8)
  EWB, Cycle 4 (n=37,27) | 7.0 (3.6) | 6.0 (4.6)
  EWB, Cycle 5 (n=29,21) | 6.3 (3.6) | 5.5 (4.7)
  EWB, Cycle 6 (n=25,20) | 6.5 (3.5) | 4.8 (3.1)
  EWB, End of Study (n=52,50) | 7.1 (4.1) | 6.0 (3.4)
  FWB, Baseline (n=56,55) | 12.3 (6.2) | 13.3 (7.4)
  FWB, Cycle 2 (n=51,41) | 12.9 (7.1) | 12.9 (7.1)
  FWB, Cycle 3 (n=41,27) | 13.0 (7.4) | 12.9 (6.9)
  FWB, Cycle 4 (n=37,26) | 12.8 (7.2) | 11.3 (7.8)
  FWB, Cycle 5 (n=29,22) | 12.7 (6.2) | 12.0 (7.6)
  FWB, Cycle 6 (n=25,20) | 11.7 (6.4) | 11.4 (6.3)
  FWB, End of Study (n=51,50) | 11.1 (7.2) | 11.5 (7.2)
  LCS, Baseline (n=56,54) | 11.0 (3.2) | 11.1 (3.8)
  LCS, Cycle 2 (n=50,45) | 10.8 (3.1) | 11.2 (3.5)
  LCS, Cycle 3 (n=42,30) | 11.0 (3.1) | 10.5 (3.2)
  LCS, Cycle 4 (n=37,27) | 11.3 (3.1) | 10.2 (3.2)
  LCS, Cycle 5 (n=28,21) | 10.8 (3.0) | 10.0 (3.9)
  LCS, Cycle 6 (n=26,20) | 10.4 (2.9) | 9.9 (4.0)
  LCS, End of Study (n=52,50) | 11.1 (3.2) | 10.8 (3.2)

9. Secondary Outcome: Changes in Quality of Life as Measured by the FACT Questionnaire
Description: The FACT Questionnaire contains 4 general and 1 lung cancer symptom-specific subscale, including PWB, SWB, EWB, FWB, and the 8-item LCS that assess symptoms commonly reported by participants with lung cancer. Each subscale was assessed by a five-point scale from 0 (not at all) to 4 (very much) to determine the quality of life. PWB, SWB and FWB scores ranged from 0-28 and EWB scores ranged from 0-24. LCS scores ranged from 0-36. For subscales of FWB and SWB, questionnaires of EWB, and additional concerns questions, the higher score represented 'Improved'. For other subscales and questionnaires, the higher score represented 'Worsened'. Missing data were replaced by the valid post-baseline assessment before. For PWB, FWB, SWB, and EWB scores and disease-specific subscale score, response of down, up or no change were defined as score changes of less than or equal to (≤)2, greater than or equal to (≥)+2, or between these values.
Time Frame: Baseline and Day 1 of Cycles 2, 3, 4, 5, 6 and End of study
Population: Safety Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 52 | 48
units on a scale
  PWB, Baseline (n=51,45) | 6.5 (3.8) | 6.0 (3.4)
  PWB, Endpoint (n=51,45) | 10.8 (5.2) | 7.8 (4.6)
  Change in PWB (n=51,45) | 4.3 (5.5) | 1.8 (4.7)
  SWB, Baseline (n=50,45) | 15.8 (6.5) | 15.4 (6.7)
  SWB, Endpoint (n=50,45) | 14.3 (7.2) | 14.4 (7.7)
  Change in SWB (n=50,45) | -1.5 (4.8) | -1.0 (6.0)
  EWB, Baseline (n=52,48) | 7.9 (3.7) | 6.2 (3.2)
  EWB, Endpoint (n=52,48) | 7.1 (4.1) | 6.0 (3.4)
  Change in EWB (n=52,48) | -0.8 (4.4) | -0.2 (4.0)
  FWB, Baseline (n=51,48) | 12.6 (6.2) | 13.4 (7.4)
  FWB, Endpoint (n=51,48) | 11.1 (7.2) | 11.7 (7.2)
  Change in FWB (n=51,48) | -1.5 (5.1) | -1.7 (6.0)
  LCS, Baseline (n=51,47) | 10.9 (3.3) | 11.2 (4.0)
  LCS, Endpoint (n=51,47) | 11.2 (3.2) | 10.7 (3.0)
  Change in LCS (n=51,47) | 0.3 (3.3) | -0.4 (4.5)
Statistical Analysis 1: Comparison: Erlotinib vs Vinorelbine; PWB, Baseline versus Endpoint; Test type: Superiority or Other; p = 0.0060, ANOVA
Statistical Analysis 2: Comparison: Erlotinib vs Vinorelbine; SWB, Baseline versus Endpoint; Test type: Superiority or Other; p = 0.6871, ANOVA
Statistical Analysis 3: Comparison: Erlotinib vs Vinorelbine; EWB Baseline versus Endpoint; Test type: Superiority or Other; p = 0.5104, ANOVA
Statistical Analysis 4: Comparison: Erlotinib vs Vinorelbine; FWB, Baseline versus Endpoint; Test type: Superiority or Other; p = 0.9927, ANOVA
Statistical Analysis 5: Comparison: Erlotinib vs Vinorelbine; LCS, Baseline versus Endpoint; Test type: Superiority or Other; p = 0.3581, ANOVA

10. Secondary Outcome: Percentage of Participants With Changes in Quality of Life as Measured by FACT Questionnaire Scores by Category of Change
Description: The FACT and the FACT-L contain 4 general and 1 lung cancer symptom-specific subscale, including PWB, SWB, EWB, FWB, and the 8-item LCS that assess symptoms commonly reported by participants with lung cancer. For subscales of FWB and SWB, questionnaires of EWB, and additional concerns questions, the higher score represented 'Improved'. For other subscales and questionnaires, the higher score represented Worsened'. For PWB, FWB, SWB, and EWB scores and disease-specific subscale score, higher scores indicated a better outcome; a response of down, up, or no change was defined as a score change of ≤ -2 (score down), ≥ +2 (score up), or between these values.
Time Frame: Baseline and End of study
Population: Safety Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 52 | 48
percentage of participants
  PWB, Score Down (n=51,45) | 7.8 | 22.2
  PWB, No Change (n=51,45) | 33.3 | 31.1
  PWB, Score Up (n=51,45) | 58.8 | 46.7
  SWB, Score Down (n=50,45) | 40.0 | 37.8
  SWB, No Change (n=50,45) | 40.0 | 40.0
  SWB, Score Up (n=50,45) | 20.0 | 22.2
  EWB, Score Down (n=52,48) | 38.5 | 33.3
  EWB, No Change (n=52,48) | 38.5 | 41.7
  EWB, Score Up (n=52,48) | 23.1 | 25.0
  FWB, Score Down (n=51,48) | 41.2 | 41.7
  FWB, No Change (n=51,48) | 33.3 | 35.4
  FWB, Score Up (n=51,48) | 25.5 | 22.9
  LCS, Score Down (n=51,47) | 17.6 | 31.9
  LCS, No Change (n=51,47) | 47.1 | 40.4
  LCS, Score Up (n=51,47) | 35.3 | 27.7

11. Secondary Outcome: Changes in Quality of Life as Assessed by FACT-L (Lung Symptoms) Questionnaire
Description: The LCS consists of 7 items of the FACT-L (3 items relating to breathing/dyspnea, and 1 item each relating to cough, weight loss, appetite, and cognition) rated on a five-point scale from 0 (not at all) to 4 (very much). The LCS total score is the sum of the scores from the 7 items. For clear thinking and good appetite, the higher score represented 'Improved'; for other subscales and questionnaires, the higher score represented 'Worsened'. Missing data were replaced by the valid post-baseline assessment before. The change of FACT-L subscore was the change from baseline to endpoint. The LCS of FACT-L is an independently validated tool that measures the disease-related symptoms of lung cancer on an overall scale of 0 (most symptomatic) to 28 (asymptomatic).
Time Frame: Baseline and Day 1 of Cycles 2, 3, 4, 5, 6 and End of study
Population: Safety Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 52 | 48
units on a scale
  Shortness of breath, Baseline (n=52,48) | 1.4 (0.7) | 1.4 (1.1)
  Shortness of breath, Endpoint (n=52,48) | 1.6 (1.0) | 1.3 (0.9)
  Shortness of breath, Change (n=52,48) | 0.2 (0.8) | -0.1 (1.2)
  Weight loss, Baseline (n=51,47) | 0.6 (0.8) | 0.8 (1.0)
  Weight loss, Endpoint (n=51,47) | 0.7 (0.9) | 0.6 (0.7)
  Weight loss, Change (n=51,47) | 0.1 (1.0) | -0.2 (1.2)
  Clear thinking, Baseline (n=52,48) | 2.4 (1.2) | 2.3 (1.3)
  Clear thinking, Endpoint (n=52,48) | 2.2 (1.3) | 2.4 (1.3)
  Clear thinking, Change (n=52,48) | -0.2 (1.1) | 0.1 (1.5)
  Coughing, Baseline (n=52,48) | 1.3 (0.6) | 1.4 (1.0)
  Coughing, Endpoint (n=52,48) | 1.4 (0.7) | 1.4 (0.8)
  Coughing, Change (n=52,48) | 0.1 (0.8) | -0.0 (1.2)
  Hair loss, Baseline (n=52,48) | 0.3 (0.6) | 0.6 (1.1)
  Hair loss, Endpoint (n=52,48) | 0.4 (0.7) | 0.4 (0.6)
  Hair loss, Change (n=52,48) | 0.1 (0.8) | -0.1 (1.2)
  Good appetite, Baseline (n=52,48) | 1.9 (0.9) | 2.0 (1.2)
  Good appetite, Endpoint (n=52,48) | 1.7 (1.1) | 1.7 (1.0)
  Good appetite, Change (n=52,48) | -0.3 (0.9) | -0.4 (1.3)
  Tightness in chest, Baseline (n=52,48) | 1.3 (0.8) | 1.2 (0.9)
  Tightness in chest, Endpoint (n=52,48) | 1.4 (0.8) | 1.3 (1.0)
  Tightness in chest, Change (n=52,48) | 0.1 (0.9) | 0.1 (1.2)
  Easy breathing, Baseline (n=52,48) | 1.7 (0.9) | 1.7 (1.1)
  Easy breathing, Endpoint (n=52,48) | 1.7 (0.9) | 1.6 (1.1)
  Easy breathing, Change (n=52,48) | -0.1 (1.1) | -0.0 (1.3)

12. Secondary Outcome: Percentage of Participants With Changes in FACT-L (Lung Symptoms) by Category of Change
Description: The LCS consists of 7 items of the FACT-L (3 items relating to breathing/dyspnea, and 1 item each relating to cough, weight loss, appetite, and cognition). The LCS total score is the sum of the scores from the 7 items, each rated on a five-point scale from 0 (not at all) to 4 (very much). For clear thinking and good appetite, the higher score represented 'Improved'; for other subscales and questionnaires, the higher score represented 'Worsened'. For each FACT-L question, the response status was defined as down, up, or no change if the score at endpoint was smaller (score down), larger than (score up), or the same as (no change) that at baseline.
Time Frame: Baseline and End of study
Population: Safety Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Number; unit: percentage of participants
Arm/Group | Erlotinib | Vinorelbine
Number analyzed (Participants) | 52 | 48
percentage of participants
  Shortness of breath, Score Down (n=52,48) | 17.3 | 18.8
  Shortness of breath, No Change (n=52,48) | 51.9 | 58.3
  Shortness of breath, Score Up (n=52,48) | 30.8 | 22.9
  Weight loss, Score Down (n=51,47) | 19.6 | 31.9
  Weight loss, No Change (n=51,47) | 51.0 | 44.7
  Weight loss, Score Up (n=51,47) | 29.4 | 23.4
  Clear thinking, Score Down (n=52,48) | 26.9 | 27.1
  Clear thinking No Change (n=52,48) | 53.8 | 43.8
  Clear thinking, Score Up (n=52,48) | 19.2 | 29.2
  Coughing, Score Down (n=52,48) | 21.2 | 22.9
  Coughing, No Change (n=52,48) | 53.8 | 50.0
  Coughing, Score Up (n=52,48) | 25.0 | 27.1
  Hair loss, Score Down (n=52,48) | 13.5 | 18.8
  Hair loss, No Change (n=52,48) | 65.4 | 60.4
  Hair loss, Score Up (n=52,48) | 21.2 | 20.8
  Good appetite, Score Down (n=52,48) | 26.9 | 35.4
  Good appetite, No Change (n=52,48) | 61.5 | 45.8
  Good appetite, Score Up (n=52,48) | 11.5 | 18.8
  Tightness in chest, Score Down (n=52,48) | 17.3 | 22.9
  Tightness in chest, No Change (n=52,48) | 55.8 | 54.2
  Tightness in chest, Score Up (n=52,48) | 26.9 | 22.9
  Easy breathing, Score Down (n=52,48) | 28.8 | 22.9
  Easy breathing, No Change (n=52,48) | 48.1 | 58.3
  Easy breathing, Score Up (n=52,48) | 23.1 | 18.8

ADVERSE EVENTS:
Time Frame: Adverse Events were monitored continuously during the study treatment and for 28 days after the last intake of study medication. Only SAE were recorded during post study treatment phase and for 28 days after the last intake of study medication.
Arm/Group | Erlotinib | Vinorelbine
Serious Adverse Events (participants affected / at risk) | 19/57 | 14/57
Other Adverse Events (participants affected / at risk) | 54/55 | 53/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=57) | Vinorelbine (N=57)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 6
Herpes zoster (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Extrapyramidal disorder (Nervous system disorders) | 1 | 0
Parkinsonism (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Alcohol withdrawal syndrome (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infarction (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Erlotinib (N=55) | Vinorelbine (N=54)
Rash (Skin and subcutaneous tissue disorders) | 38 | 3
Diarrhoea (Gastrointestinal disorders) | 20 | 7
Mouth ulceration (Gastrointestinal disorders) | 9 | 1
Constipation (Gastrointestinal disorders) | 7 | 7
Mucosal inflammation (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Insomnia (Psychiatric disorders) | 5 | 7
Vomiting (Gastrointestinal disorders) | 4 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Anaemia (Blood and lymphatic system disorders) | 3 | 1
Conjunctivitis (Infections and infestations) | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4
Nausea (Gastrointestinal disorders) | 3 | 5
Stomatitis (Gastrointestinal disorders) | 3 | 4
Tinea cruris (Infections and infestations) | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Hypertension (Vascular disorders) | 3 | 0
Abdominal distension (Gastrointestinal disorders) | 2 | 4
Pyrexia (General disorders) | 3 | 8
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Fatigue (General disorders) | 1 | 6
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 0
Oedema (General disorders) | 3 | 4
Folliculitis (Infections and infestations) | 4 | 0
Decreased appetite (Metabolism and nutrition disorders) | 16 | 24
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Headache (Nervous system disorders) | 3 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.